CLINICAL TRIAL: NCT07185269
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase Ib/II Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Immunogenicity of Anti-BDCA2 Antibody SSGJ-626 in Subjects With Systemic Lupus Erythematosus
Brief Title: The Purpose of This Study is to Evaluate the Efficacy and Safety of 626 in the Treatment of SLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-626-SLE-Ib/II-01
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group M1 (Experimental): dose level 1 of 626
  Interventions: Drug: 626; Drug: Placebo
- Group M2 (Experimental): dose level 2 of 626
  Interventions: Drug: 626; Drug: Placebo
- Group M3 (Experimental): dose level 3 of 626
  Interventions: Drug: 626; Drug: Placebo
- Group M4 (Experimental): dose level 4 of 626
  Interventions: Drug: 626; Drug: Placebo
- 626 Dose A (Experimental): 626 Dose A subcutaneous (SC) injection.
  Interventions: Drug: 626
- 626 Dose B (Experimental): 626 Dose B subcutaneous (SC) injection
  Interventions: Drug: 626
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 626 — 626 subcutaneous (SC) injection. Placebo subcutaneous (SC) injection.
  Arms: Group M1; Group M2; Group M3; Group M4
Drug: 626 — 626 subcutaneous (SC) injection.
  Arms: 626 Dose A; 626 Dose B
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Group M1; Group M2; Group M3; Group M4; Placebo

SUMMARY:
This study will evaluate the effect and safety of 626 in patients with SLE

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease with heterogeneous manifestations and disease course. Despite advances in medical care, there are still significant unmet needs in SLE with persistent disease activity, disease flares, intolerance to standard of care (SOC) therapies, and development of organ damage and co-morbidities.

The purpose of this study is to demonstrate the clinical efficacy and safety of 626 added to standard of care (SoC) therapy compared to placebo with SoC therapy in subjects with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand protocol requirements and sign a written ICF.
* Male or female subjects aged 18-70 years when signing the ICF.
* Body weight between 40 and 90 kg.
* Diagnosed with SLE at least 6 months before the Screening Visit by a qualified physician，confirmed according to the 2019 SLE European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE.
* At screening, meet at least one of the following criteria:

  1. Anti-nuclear antibody (ANA) titer ≥ 1:80;
  2. Positive anti-dsDNA antibody..
* Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≥6 with clinical SLEDAI score ≥4 points at Screening and Baseline Visit .
* Currently receiving at least one of the SOC SLE medications: oral corticosteroid, antimalarial and/or immunosuppressive agent.

Exclusion Criteria:

* Study participant has a mixed connective tissue disease, and/or overlap syndrome of systemic lupus erythematosus (SLE) with systemic sclerosis.
* Study participant has any medical or psychiatric condition (including conditions due to neuropsychiatric SLE) that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study. This includes study participants with a life-threatening condition
* Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
* History of cancer.
* Active severe lupus nephritis present within 2 months prior to baseline. Or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2, or protein:creatinine ratio >2.0 g/g.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-08-12 (Estimated); Study Completion 2028-11-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | During the 32- or 36-week study period
  Incidence of adverse events will be summarized by SOC and PT for each treatment group, and also be summarized by severity and association with the study treatments.

SECONDARY OUTCOMES:
SLE Responder Index (SRI-4) | During the 20- or 24-week treatment period
  Proportion of subjects achieving an SLE Responder Index (SRI-4) response
BILAG-based Combined Lupus Assessment (BICLA) Response | During the 20- or 24-week treatment period
  Proportion of patients achieving a BILAG-based Combined Lupus Assessment (BICLA) response

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) | During the 32- or 36-week study period
Area under the Concentration-Time Curve up to the Last Measurable Concentration（AUC0-last） | During the 32- or 36-week study period
Time to Peak Concentration（Tmax ） | During the 32- or 36-week study period

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No